CLINICAL TRIAL: NCT00654342
Title: Comparison Between ex Vivo and in Vivo Injection of Blue Dye in Sentinel Lymph Node Mapping for Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University (Other)
Responsible Party: Department of Surgery, colleage of medicine,, Chung-Ang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: caugs_01
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2008-04

CONDITIONS: Sentinel Lymph Node Biopsy; Colon Cancer
Keywords: Sentinel lymph node-colon cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Postoperative Period

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): In vivo injection group
  Interventions: Procedure: Intraoperative injection (in vivo)
- 2 (Other): Ex vivo injection group
  Interventions: Procedure: Postoperative injection (ex vivo)

INTERVENTIONS:
Procedure: Intraoperative injection (in vivo) — Intraoperative injection
  Arms: 1
Procedure: Postoperative injection (ex vivo) — postoperative injection
  Arms: 2

SUMMARY:
The technique of sentinel lymph node mapping in patients with colon cancer varies among reports, and the optimal method remain to be established. The purpose of this study was to determine the optimal injection technique for sentinel lymph node mapping for colon cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage I - III colon cancer patients

Exclusion Criteria:

* cancer located at the low rectum which were located within 10 cm of the dentate, recurrent or metastatic colon carcinoma, adjacent organ invasion tumor, prior chemotherapy or radiation, cancer with intestinal obstruction, past intestinal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy & sensitivity of sentinel lymph node mapping | After confirmed pathological report

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Chung-Ang university Hospital, Seoul, South Korea